CLINICAL TRIAL: NCT00869531
Title: Healthgrain WP 4.4.3: Effects of Whole Grain on Weight Maintenance/Weight Reduction in Overweight Subjects
Brief Title: Effect of Wholegrain Wheat on Body Weight and Composition and Cardiovascular Risk
Acronym: HEALTHGRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: BARILLA G. e R. Fratelli S.p.A., Parma, Italy (Unknown); European Commission (Other)
Responsible Party: Arne Astrup, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B223
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Obesity
Keywords: Obesity; wholegrain; wheat; cardiovascular disease
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WW (Experimental): wholegrain wheat
  Interventions: Other: wholegrain
- RW (Active Comparator): refined wheat
  Interventions: Other: refined wheat

INTERVENTIONS:
Other: wholegrain — wholegrain wheat vs. refined wheat products
  Arms: WW
Other: refined wheat — refined wheat products
  Arms: RW

SUMMARY:
The aim of this study is to investigate the potential beneficial effect of wholegrain on body weight and composition as well as cardiovascular risk in overweight women.

DETAILED DESCRIPTION:
Objective: To study the effect of the 'wholegrain concept', i.e. high intake of wheat wholegrain (WW) vs. refined wheat (RW) grain products on body weight and composition.

Design: In this open-labeled randomized trial, 72 postmenopausal women with metabolic syndrome features were prescribed a mild calorie-restricted diet with a deficit of ~1,250kJ/d. Following 2 weeks run-in period on RW products, they were randomized to 12 weeks intervention with RW or WW products providing 2,000kJ/d.

ELIGIBILITY:
Inclusion Criteria:

* BMI 27-37
* Postmenopausal (>1y) women
* 40-70 years old

Exclusion Criteria:

* Medication (hypertensive treatment not included)
* BP > 160/100
* Fasting glucose > 7mM
* Fasting cholesterol > 6.5mM
* Smoking
* Known chronic illnesses

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Body weight and composition | 0, 6 and 12 wks

SECONDARY OUTCOMES:
Cardiovascular risk markers | 0, 6 and 12 wks
Fecal parameters | 0 and 12 wks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department og Human Nutrition, Frederiksberg C, Denmark

REFERENCES:
- See also: EU project homepage — http://www.healthgrain.org